CLINICAL TRIAL: NCT05472779
Title: Periurethral vs Intravaginal Estrogen for Prevention of Recurrent Urinary Tract Infections: TAPER (Techniques of APplying Vaginal Estrogen for Prevention of Recurrent Urinary Tract Infections) Trial
Brief Title: Periurethral vs Intravaginal Estrogen for Prevention of Recurrent Urinary Tract Infections
Acronym: TAPER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stephanie Wang Zuo (Other)
Responsible Party: Sponsor-Investigator, Stephanie Wang Zuo, Adjunct Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY22010147
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-12

CONDITIONS: Recurrent Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravaginal Estrogen Application (Active Comparator): Intravaginal application of 1 gram estradiol cream at bedtime twice a week for 6 months
  Interventions: Drug: Intravaginal application of estradiol cream
- Periurethral Estrogen Application (Experimental): Periurethral application of 0.5 gram estradiol cream at bedtime twice a week for 6 months
  Interventions: Drug: Periurethral application of estradiol cream

INTERVENTIONS:
Drug: Periurethral application of estradiol cream — The experimental group will apply estradiol cream in a different location (periurethral) and at a smaller dose (0.5 gram) compared to the control group.
  Arms: Periurethral Estrogen Application
Drug: Intravaginal application of estradiol cream — The control group will apply 1 gram estradiol cream intravaginally using an applicator.
  Arms: Intravaginal Estrogen Application

SUMMARY:
Due to rising antibiotic resistance, there has been a focus on non-antibiotic prophylactic measures for postmenopausal patients with recurrent urinary tract infections (rUTI), one of which is the safe and efficacious option of vaginal estrogen therapy. Standard application of vaginal estrogen cream entails intravaginal application of the cream twice a week, but some providers counsel patients with rUTI to apply a small, pea-sized amount to the periurethral area. This ideally reduces the amount of vaginal estrogen used while attaining a similar effect. However, to date, there is no data to prove that the periurethral technique of application is similar or non-inferior to intravaginal application in preventing UTI.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (definition: No menses for 1 or more years or surgical menopause (bilateral oophorectomy). If there is a past history of hysterectomy, patient must be age 56 or older (95th percentile for age at menopause) or have laboratory evidence of menopause (ie. FSH >30)
* Meets criteria for recurrent urinary tract infections (UTIs) with 2 or more UTI in 6 months or 3 or more UTI in 1 year
* May include patients who used vaginal estrogen previously if they have stopped use for 3 or more months prior to inclusion into study.
* Patients must be recommended vaginal estrogen as part of normal clinical care for prevention of recurrent UTI

Exclusion Criteria:

* Current use of vaginal or oral estrogen products
* Inability or refusal to use vaginal estrogen
* Daily antibiotic use
* Significant vaginal stenosis (eg. due to lichen sclerosis, radiation or obliterative prolapse surgery) that would prohibit use of a vaginal applicator (ie. genital hiatus <1cm)
* Inability to use vaginal applicator and without caregiver who can administer (eg. provider-managed pessary use, significant arthritis)
* Frequent (1x weekly or more frequent) use of bladder instillations containing an antibiotic
* Known hydronephrosis as a result of incomplete bladder emptying
* Use of intermittent or indwelling urinary catheterization
* Known bladder stones, mesh erosion into bladder, or foreign object in bladder
* Unable to consent for self
* Active treatment for an estrogen-dependent malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who are UTI-free at 6 months | 6 months

SECONDARY OUTCOMES:
Change from baseline in urinary symptoms at 6 months | Baseline, 6 months
  Questionnaire assessment of urinary symptoms and symptom distress (Urogenital Distress Inventory, Short Form), total score range 0-100 with higher numbers representing worse urinary symptoms
Change from baseline in vaginal symptoms at 6 months | Baseline, 6 months
  Questionnaire assessment of vaginal symptoms and bother using 5-point Likert scale, developed by research team
Change from baseline in sexual function at 6 months | Baseline, 6 months
  Questionnaire assessment of sexual function (Female Sexual Function Index-6) with scores ranging from 2 to 30, with 19 and below denoting sexual dysfunction.
Amount of estrogen cream used | 6 months
  Estradiol cream tubes will be weighed at each research visit in grams
Participant experience with use of estrogen cream | 6 months
  Questionnaire assessment of patient experience using 5-point Likert and open-ended questions, developed by the research team
Change from baseline in vaginal pH at 6 months | Baseline, 6 months
  Assessment using pH strips during pelvic examination
Change from baseline in vaginal maturation index at 6 months | Baseline, 6 months
  Assessment of vaginal cell types using a superficial swab, collected from proximal vagina
Change from baseline in Vaginal and urinary Lactobacillus levels at 6 months | Baseline, 6 months
  Clean catch urine and vaginal swab sample collection with quantification of Lactobacillus
Change from baseline in Vaginal and urinary E. coli levels at 6 months | Baseline, 6 months
  Clean catch urine and vaginal swab sample collection for quantification of E. coli

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie W Zuo, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (4):
- United States (4):
  - UPMC Lemieux Sports Complex, Cranberry Township, Pennsylvania
  - UPMC Hamot, Erie, Pennsylvania
  - University of Pittsburgh Medical Center-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Passavant-McCandless, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No